CLINICAL TRIAL: NCT00015691
Title: A Randomized, Double-Blind, Placebo-Controlled Study of Metformin and Rosiglitazone, Alone or in Combination, in HIV-Infected Subjects With Hyperinsulinemia and Elevated Waist/Hip Ratio
Brief Title: Metformin and Rosiglitazone, Alone or in Combination, in HIV-Infected Patients With Insulin and Fat Abnormalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: A5082; AACTG A5082; ACTG A5082; 10913 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2001-05-01; First posted 2001-08-31 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections; Lipodystrophy; Hyperinsulinemia
Keywords: Drug Therapy, Combination; Adipose Tissue; Area Under Curve; Hypoglycemic Agents; Anthropometry; Hyperinsulinemia; Metformin; BRL 49653; Insulin; Glucose Tolerance Test
MeSH Terms: conditions — HIV Infections; Lipodystrophy; Hyperinsulinism; Insulin Resistance | interventions — Metformin; Rosiglitazone

INTERVENTIONS:
Drug: Metformin hydrochloride
Drug: Rosiglitazone maleate

SUMMARY:
The purpose of this study is to see whether metformin alone, rosiglitazone alone, or metformin and rosiglitazone together will lower insulin levels in the blood and decrease fat in the abdomen or other parts of the body.

Studies have shown that certain anti-HIV medications can cause a number of side effects, including high blood sugar (resulting from the body's failure to use insulin), high insulin, and excess fat build-up in the abdominal area. These side effects are known to increase the risk of heart disease. Metformin and rosiglitazone are 2 drugs that have been shown to lower insulin resistance and lessen abdominal fat in patients who are not HIV-infected. This study will investigate the use of these drugs in HIV-infected patients.

DETAILED DESCRIPTION:
Recent studies have documented hyperglycemia, insulin resistance, and glucose intolerance in a seemingly increasing proportion of patients with HIV infection. Other studies have described a variety of syndromes of fat accumulation and fat loss, including abdominal obesity. Although initially attributed specifically to protease inhibitors (PI), these abnormalities also have been observed in antiretroviral-experienced but PI-naive patients. Hyperinsulinemia and abdominal obesity are strong independent risk factors for coronary artery disease. In noninfected patients, metformin and thiazolidinediones have been shown to reduce insulin resistance by different mechanisms and also to reduce visceral adiposity. This study investigates the use of metformin and rosiglitazone, a member of the thiazolidinedione class, in HIV-infected patients with hyperinsulinemia and central fat accumulation.

At study entry, clinical and laboratory assessments are performed. A standard OGTT, with plasma samples drawn over 120 minutes, will be performed for glucose and insulin determinations. After completion of entry evaluations, patients are assigned randomly to 1 of 4 double-blinded treatment arms:

Arm A: Metformin plus rosiglitazone placebo. Arm B: Metformin placebo plus rosiglitazone. Arm C: Metformin plus rosiglitazone. Arm D: Metformin placebo plus rosiglitazone placebo. Patients who are still on study drugs at Week 16 (at either full or reduced dose) are switched to the open-label phase to receive the combination of metformin and rosiglitazone through Week 32. Patients have evaluations at Weeks 2, 4, 8, 12, 16, 18, 20, 24, 28, and 32. [AS PER AMENDMENT 02/05/02: Evaluations must be performed under fasting conditions.] Safety indices, fasting insulin and glucose levels, visceral [AS PER AMENDMENT 02/05/02: and subcutaneous abdominal] fat are assessed. [AS PER AMENDMENT 02/05/02: Patients who discontinue study treatment due to pregnancy during the study will have the Week 32 evaluations (except CT and DEXA scans).] [AS PER AMENDMENT 02/05/02: A mid-thigh measurement was added to the study as a secondary endpoint to look for changes in extremity subcutaneous fat from therapy with rosiglitazone. Rosiglitazone and other peroxisome proliferator-activated receptor (PPAR) gamma activators increase subcutaneous adipogenesis and may thus increase subcutaneous fat and improve insulin resistance in this way.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have a viral load (level of HIV in the blood) below 10,000 copies/ml, within 30 days before study entry.
* Have a fasting blood insulin level at 15 micro IU/ml or greater; or a 2-hour insulin at least 75 micro IU/ml or greater following 75 g glucose load; or a 2-hour glucose greater than 140 mg/dl following 75 g glucose load AND fasting serum insulin at least 10 micro IU/ml or greater, within 30 days before study entry.
* Meet physical restrictions based on the amount and location of body fat and also on height and weight.
* Have noticed changes in the location of their body fat during the course of their HIV disease.
* Are 18 to 65 years old.
* Have taken the same anti-HIV drugs for at least 60 days before study entry and do not plan to change these drugs for the entire study.
* If taking hormones, have been on the same treatment for at least 6 months before study entry and do not plan to change for the entire study. Hormones include birth control pills, estrogen, or progestin for women and testosterone for men. If hormones were taken and then stopped, the treatment must have ended at least 6 months before the patient enters the study.
* Have a negative pregnancy test within 30 days before taking the study drugs, if female and able to have children.
* Agree to avoid trying to become pregnant or causing someone to become pregnant. Agree not to donate sperm or participate in other fertilization procedures. If sexually active, agree to use [AS PER AMENDMENT 02/05/02: 1] effective method of birth control while taking the study medications and for at least 30 days after stopping the study medications. Women who are not able to give birth or whose male partner is sterile are not required to use birth control.
* Several changes have been made to this study. In earlier versions, a fasting blood insulin above 15 micro IU/ml was the only level accepted. Now there are several other insulin/glucose levels included. In addition, the timing of pregnancy tests has changed from 14 days to 30 days.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are allergic to metformin or rosiglitazone.
* Are pregnant or breast-feeding.
* Abuse drugs or alcohol.
* Have diarrhea, nausea, or vomiting.
* Have heart disease.
* Are taking or have taken drugs to control blood sugar.
* Have taken any of the following drugs within 6 months before study entry: high-dose estrogen, high-dose testosterone, high-dose testosterone gel, testosterone creams, growth hormone, steroids to increase body size, DHEA or androstenedione (sold over the counter), prednisone and other steroid drugs at high doses, drugs to increase appetite, experimental drugs to increase appetite or weight gain, drugs that affect the immune system, pentoxifylline, thalidomide, niacin (a multivitamin containing niacin is okay), hydroxyurea, and cimetidine.
* Are taking ritonavir with simvastatin or lovastatin (drugs to lower cholesterol).
* Are taking drugs not approved by the FDA or of unknown identity, in experimental studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105
Dates: Primary Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Mulligan, Study Chair; Steven Grinspoon, Study Chair
Locations (34):
- United States (34):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Willow Clinic, Menlo Park, California
  - Univ of California, San Diego, San Diego, California
  - Univ of California San Francisco, San Francisco, California
  - San Mateo AIDS Program / Stanford Univ, Stanford, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Hawaii, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Univ of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Washington Univ / St Louis Connect Care, St Louis, Missouri
  - Washington Univ School of Medicine, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Hadigan C, Rabe J, Grinspoon S. Sustained benefits of metformin therapy on markers of cardiovascular risk in human immunodeficiency virus-infected patients with fat redistribution and insulin resistance. J Clin Endocrinol Metab. 2002 Oct;87(10):4611-5. doi: 10.1210/jc.2002-020709. PMID 12364443